CLINICAL TRIAL: NCT00249652
Title: Drug Treatment for Transplant Candidates
Brief Title: Transplant and Addiction Project (TAP) - 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15772-1; R01-15772-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: End Stage Liver Disease; End Stage Renal Disease; Substance-Related Disorders
Keywords: End stage liver disease; End stage renal disease; Substance-Related Disorders
MeSH Terms: conditions — End Stage Liver Disease; Kidney Failure, Chronic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP (Experimental): MI-based phone intervention.
  Interventions: Behavioral: TAP
- TAU (Other): Treatment As Usual
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: TAP — 12-session motivational interviewing-based telephone intervention.
  Arms: TAP
Other: TAU — The usual care group will receive the same medical services they would otherwise receive if they were not in this study.
  Arms: TAU

SUMMARY:
The purpose of this study is to test a novel distance-based (telephone) intervention to help transplant candidates with current or recent substance abuse to stay "clean and sober" both prior and following transplant surgery.

DETAILED DESCRIPTION:
Participants who need a liver or renal transplant and who are ineligible due to current or recent (past 6 months) alcohol and/or other drug abuse are being recruited from the transplant programs at St. Luke's-Roosevelt Hospital Center (renal), Columbia Presbyterian Hospital (renal/liver) and Virginia Commonwealth University Medical Center (liver). Baseline and follow-up computer-assisted assessments and structured clinical interviews along with collection of biological samples (urine, hair) will occur in the transplant clinics; however, phone counseling sessions originate at St. Luke's. Participants are randomly assigned to one of two treatments: (1) usual care (no phone counseling) or (2) usual care + counseling. The telephone counseling sessions are designed to help participants become motivated to remain abstinent and improve other health behaviors such as sleep or stress management.

ELIGIBILITY:
Inclusion Criteria:

* End stage liver or renal disease
* Having used drugs or alcohol during the past 6 months
* Turned down for transplant due to current or recent substance use
* Access to telephone

Exclusion Criteria:

* Psychotic or other unstable serious psychiatric disorders that preclude full, active participation
* Moderate to severe hepatic encephalopathy
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-09; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Abstinence | 3 month time frame

SECONDARY OUTCOMES:
Stage of Change, illness response, psychological stress | 3 month time frame

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Haller, Principal Investigator — St. Luke's Roosevelt Hosp Cntr (New York)
Locations (3):
- United States (3):
  - Behavioral Science Research Unit, New York, New York
  - Renal & Islet Transplant, Center for Liver Disease, New York, New York
  - Liver Transplant Program, Richmond, Virginia

REFERENCES:
- [Background] Wagner CC, Haller DL, Olbrisch ME. Relapse prevention treatment for liver transplant patients. J Clin Psychol Med Settings. 1996 Dec;3(4):387-98. doi: 10.1007/BF01994021. PMID 24226847
- [Background] Presented at the Ninth Annual International Liver Transplantation Society Congress, Barcelona, Spain, June 2003.